CLINICAL TRIAL: NCT01391312
Title: A Pilot Study of BOTOX® Cosmetic in the Treatment of Moderate to Severe Glabellar Lines - Establishing Patient Satisfaction
Brief Title: Patient Satisfaction Study of BOTOX® Cosmetic in the Treatment of Moderate to Severe Frown Lines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GMA-BTXC-11-001
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-08

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- botulinum toxin Type A (Active Comparator): Botulinum toxin Type A 20U (total dose) injected into the glabellar region on Day 0.
  Interventions: Biological: botulinum toxin Type A
- placebo (Normal Saline) (Placebo Comparator): Normal Saline (placebo) injected into the glabellar region on Day 0.
  Interventions: Drug: normal saline (placebo)

INTERVENTIONS:
Biological: botulinum toxin Type A — botulinum toxin Type A 20U (total dose) injected into the glabellar region on Day 0.
  Other Names: BOTOX® Cosmetic, Vistabel®, Vistabax®
  Arms: botulinum toxin Type A
Drug: normal saline (placebo) — Normal saline (placebo) injected into the glabellar region on Day 0.
  Arms: placebo (Normal Saline)

SUMMARY:
This was a pilot study to observe patient satisfaction with BOTOX® Cosmetic treatment in glabellar rhytides (frown lines) using a new treatment satisfaction measure.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe glabellar wrinkles (frown lines)

Exclusion Criteria:

* Previous treatment with botulinum toxin therapy of any serotype
* Facial non-ablative resurfacing laser or light treatment, microdermabrasion, or superficial peels within 3 months
* Any facial cosmetic procedure with medium depth to deep facial chemical peels (e.g., trichloroacetic acid and phenol), mid-facial or periorbital laser skin resurfacing or permanent make-up within 6 months
* Mid-facial or periorbital treatment with non-permanent soft tissue fillers
* Subjects planning a facial cosmetic procedure or visible scars
* Previous cosmetic surgery to the upper face(e.g., prior periorbital surgery, facial lift, brow lift, eyelid lift or eyebrow surgery)
* Diagnoses of Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis
* History of facial nerve palsy
* A planned extended absence during the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- East Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age Continuous [Mean (Standard Deviation); unit: Years] | 46.3 (12.8) | 54.5 (7.1) | 50.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Improvement in Subject Global Assessment of Change at Day 30
Description: Subjects assessed the improvement of their glabellar lines (area between the eyebrows) by answering the question: Compared to before receiving the study treatment, How do you currently feel about the appearance of your glabellar lines? on a 7-point scale where 0=Very much improved, 1=Much improved, 2=Minimally improved, 3=No change, 4=Minimally worse, 5=Much worse, 6=Very much worse. Improvement was defined as responses: 0=Very much improved, 1=Much improved and 2=Minimally improved.
Time Frame: Day 30
Population: Participants from the Intent-to-treat population (all randomized participants) with data available for the time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 20
Percentage of participants | 94.7 (0.84) | 0.00 (0.00)

2. Secondary Outcome: Percentage of Facial Wrinkle Scale Responders at Maximum Attempted Muscle Contraction at Day 30
Description: The Investigator rated the subject's severity of glabellar lines (between the eyebrows) at maximum attempted muscle contraction using the 4-point Facial Wrinkle scale where 0=None (Best), 1=Mild, 2=Moderate, 3=Severe (Worse) at day 30. Responders were defined as participants with a score of 0=None or 1=Mild.
Time Frame: Day 30
Population: Participants from the Intent-to-treat population (all randomized participants) with data available for the time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 19 | 20
Percentage of participants | 100 | 10

3. Secondary Outcome: Percentage of Facial Wrinkle Scale Responders at Maximum Attempted Muscle Contraction at Day 60
Description: The Investigator rated the subject's severity of glabellar lines (between the eyebrows) at maximum attempted muscle contraction using the 4-point Facial Wrinkle scale where 0=None (Best), 1=Mild, 2=Moderate, 3=Severe (Worse) at day 60. Responders were defined as participants with a score of 0=None or 1=Mild.
Time Frame: Day 60
Population: Participants from the Intent-to-treat population (all randomized participants) with data available for the time-point.
Measure: Number; unit: Percentage of participants
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 18 | 19
Percentage of participants | 77.8 | 5.3

ADVERSE EVENTS:
Description: Serious adverse events and adverse events were assessed in all participants with at least 1 post-baseline assessment.
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 2/19 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=19) | Placebo (Normal Saline) (N=20)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Very small bruise (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.